CLINICAL TRIAL: NCT00019994
Title: Immunization of Patients With Metastatic Melanoma Using a Class II Restricted Peptide From the GP100 Antigen and Class I Restricted Peptides From the GP100 and MART-1 Antigens
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067391; NCI-99-C-0159; NCI-T99-0079; NCT00001833 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2003-03

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; aldesleukin; incomplete Freund's adjuvant

INTERVENTIONS:
Biological: MART-1 antigen
Biological: aldesleukin
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of vaccine therapy in treating patients who have metastatic melanoma that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the clinical response to immunization using gp100:44-59 antigen peptide plus gp100:209-217 (210M) and MART-1:26-35 (27L) antigen peptides in patients with metastatic melanoma who are HLA-DRB1*0401 and HLA-A0201 positive.
* Determine the clinical response to immunization using gp100:44-59 antigen peptide alone in patients with metastatic melanoma who are HLA-DRB1*0401 positive but HLA-A0201 negative.
* Determine the immunologic response in patients treated with these regimens as measured by changes in T-cell precursors from before to after treatment.
* Evaluate the toxicity profiles of these regimens in these patients.

OUTLINE: Patients are assigned to one of three immunization groups based on HLA-A0201 status and prior gp100:209-217 (210M) antigen peptide immunization:

* Group 1 (HLA-A0201 positive and no prior gp100:209-217 [210M] antigen peptide): Patients receive gp100:44-59 and gp100:209-217 (210M) antigen peptides emulsified together in Montanide ISA-51 (ISA-51) subcutaneously (SC) and gp100:44-59 and MART-1:26-35 (27L) antigen peptides emulsified together in ISA-51 SC.
* Group 2 (HLA-A0201 positive and prior gp100:209-217 [210M] antigen peptide): Patients receive treatment as in group 1.
* Group 3 (HLA-A0201 negative and no prior gp100:209-217 [210M] antigen peptide): Patients receive gp100:44-59 antigen peptide emulsified in ISA-51 SC alone.
* All groups: Treatment repeats every 3 weeks for 4 doses in the absence of disease progression or unacceptable toxicity. Patients with complete response after 4 doses receive a maximum of 2 additional doses. Patients with stable disease or minor, mixed, or partial response after 4 doses receive a maximum of 12 additional doses. Patients with no response after 4 doses receive immunization with the same peptides and interleukin-2 IV over 15 minutes every 8 hours for a maximum of 12 doses beginning 1 day after each immunization.

Patients are followed at 3-4 weeks.

PROJECTED ACCRUAL: A total of 45-75 patients (15-25 per immunization group) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven metastatic melanoma that has failed standard treatment
* HLA-DRB1*0401 positive
* Known HLA-A0201 status

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 90,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 mg/dL
* AST or ALT less than 3 times normal
* Hepatitis B surface antigen negative

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No symptomatic cardiac disease

Immunologic:

* No autoimmune disease
* No primary or secondary immunodeficiency disease
* HIV negative

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active systemic infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunization to the entire gp100 molecule
* At least 3 weeks since prior gp100:209-217 antigen peptide
* At least 3 weeks since other prior biologic therapy

Chemotherapy:

* At least 3 weeks since prior chemotherapy

Endocrine therapy:

* At least 3 weeks since prior endocrine therapy
* No concurrent steroid therapy

Radiotherapy:

* At least 3 weeks since prior radiotherapy

Surgery:

* Prior surgery for cancer allowed

Other:

* At least 3 weeks since any prior therapy except surgery for cancer

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-10; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Background] Phan GQ, Touloukian CE, Yang JC, Restifo NP, Sherry RM, Hwu P, Topalian SL, Schwartzentruber DJ, Seipp CA, Freezer LJ, Morton KE, Mavroukakis SA, White DE, Rosenberg SA. Immunization of patients with metastatic melanoma using both class I- and class II-restricted peptides from melanoma-associated antigens. J Immunother. 2003 Jul-Aug;26(4):349-56. doi: 10.1097/00002371-200307000-00007. PMID 12843797